CLINICAL TRIAL: NCT00323544
Title: A Phase 3, Open Label, Randomised, Parallel Group Study to Compare the Effect on Prevention and Resolution of Treatment Related Adverse Events of a Simplified, Once Daily Regimen of a Fixed Dose Combination Tablet of Emtricitabine and Tenofovir DF Versus Twice Daily co-Formulated Zidovudine and Lamivudine (Combivir®) or Zidovudine and Lamivudine, in Virologically Suppressed, HIV Infected Patients Taking Efavirenz
Brief Title: SWEET: Once Daily Truvada Versus Twice Daily Combivir for the Treatment of HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Cham Herath, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-MC-164-0111
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV 1; HIV 1 infection
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Lamivudine; lamivudine, zidovudine drug combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: zidovudine and lamivudine (Combivir®)
Drug: emtricitabine and tenofovir DF

SUMMARY:
This study will investigate whether the simplified regimen of a once daily fixed dose combination of Truvada (emtricitabine and tenofovir disoproxil fumarate [DF]) will be associated with a reduced rate of adverse events, seen with long term use of antiretrovirals, as well as improved adherence compared to a twice daily fixed dose combination of Combivir.

DETAILED DESCRIPTION:
The success of HAART is largely dependant on an individual's ability to adhere strictly to an antiretroviral regimen. Regimen characteristics that affect adherence include dosing frequency and pill burden. Several studies have shown improved adherence with lower pill burden and a meta-analysis of the virological outcome in relation to pill burden has shown a significant correlation between lower pill burden and better virological outcome. A systematic review of studies across a range of medical specialties demonstrated that once daily therapy improves adherence relative to more frequent dosing although statistical significance was not demonstrated relative to twice daily regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged > 18 years.
2. HIV positive.
3. Stable antiretroviral therapy consisting of efavirenz (EFV) given with Combivir® or zidovudine (AZT) + lamivudine (3TC) for at least 6 months.
4. Patients with viral loads < 50 copies/ml on last 2 consecutive tests and < 400 copies/ml for > 3 months.
5. Patients requiring a lipid lowering agent must be established on a stable dose/frequency for at least 12 weeks prior to Baseline and be expected to continue on stable dose/frequency for the duration of the study.
6. Negative serum pregnancy test (females of childbearing potential only).
7. Willingness to use effective contraception (such as barrier or coil methods) by both males and females while on study treatment and for 30 days following study drug completion.
8. The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

1. Pregnant or lactating female.
2. History of AZT monotherapy.
3. Use of anabolic steroids, with the exception of testosterone for documented hypogonadism, within 90 days prior to the Baseline visit.
4. Documented parvovirus infection.
5. Use of erythropoietin within the last six weeks.
6. Patients who have had a blood transfusion in the last six weeks.
7. Karnofsky score < 50.
8. Prior history of significant renal disease.
9. Prior history of osteopenia/osteoporosis.
10. Creatinine clearance < 60mL/min.
11. AST/ALT > 5 x upper limits of normal (ULN).
12. Previous adefovir dipivoxil or cidofovir therapy.
13. Known history of resistance (including primary resistance) to any of the study medications - tenofovir disoproxil fumarate (TDF), emtricitabine (FTC), AZT, 3TC, or EFV.
14. Patients receiving ongoing therapy with any of the following (administration of any of the following medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period):

    * Nephrotoxic agents
    * Probenecid
    * Systemic chemotherapeutic agents (i.e. cancer treatment medications)
    * Systemic corticosteroids
    * Interleukin 2 (IL 2)
    * Drugs that interact with efavirenz
    * Dihydroergotamine
    * Ergotamine
    * Midazolam
    * Triazolam
    * Cisapride
    * Rifampin
    * Ergonovine
    * Methylergonovine
15. Patients with known hypersensitivity to any of the study medications or excipients.
16. Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic therapy within 15 days prior to Screening.
17. Patients who are currently taking part in any other clinical trial or have taken part in a clinical trial of a new chemical entity within 1 month prior to Screening.
18. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the dosing requirements.
19. Patients with cancer (except basal cell carcinoma).
20. Co-infection with hepatitis B virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the study is a change from baseline in absolute haemoglobin at Week 24.

SECONDARY OUTCOMES:
The secondary endpoints in this study include: Change from baseline in absolute haemoglobin at Week 48
Lipids profile: change from baseline in total cholesterol (TC), low density lipoprotein (LDL), high density lipoprotein (HDL), TC/HDL, and triglyceride (TG)
Quality of life (QoL)
Measures of treatment adherence (Medication Adherence Self-Report Survey [MASRI] questionnaire)
Measures of regimen intrusiveness (HIS and Brief Medication Questionnaire [BMQ])
Changes in markers of body composition from dual energy x-ray absorptiometry (DEXA) scans (a sub-study)
HIV RNA: proportion of patients with HIV ribonucleic acid (RNA) < 400 copies/mL; proportion of patients with HIV RNA < 50 copies/mL and change from baseline in log10 copies/mL at Weeks 24 and 48
CD4: change from baseline in CD4 counts
Treatment adherence and acceptability
Use of lipid lowering drugs (number of patients and duration of use)
Adverse events (AEs): AEs will be coded and the coded terms will be used to summarize the count of patients with any event, intensity of each event (highest intensity will be used if an event is reported more than once by a patient) and relationship to:
Other lab tests: results at baseline and changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Avila, MD, Study Director — Gilead Sciences, Ltd.
Locations (1):
- Gilead Sciences, Cambridge, United Kingdom

REFERENCES:
- [Derived] Fisher M, Moyle GJ, Shahmanesh M, Orkin C, Kingston M, Wilkins E, Ewan J, Liu H, Ebrahimi R, Reilly G; SWEET (Simplification With Easier Emtricitabine Tenofovir) group UK. A randomized comparative trial of continued zidovudine/lamivudine or replacement with tenofovir disoproxil fumarate/emtricitabine in efavirenz-treated HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):562-8. doi: 10.1097/QAI.0b013e3181ae2eb9. PMID 19561519
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-MC-164-011_Synopsis_Public%20Disclosure_Final.pdf